CLINICAL TRIAL: NCT00929175
Title: Antihypertensive Effect of Continuous Positive Airway Pressure (CPAP) in Resistant Hypertensive Patients With Sleep Apnea: Randomized Clinical Trial
Brief Title: Antihypertensive Effect of Continuous Positive Airway Pressure in Resistant Hypertensive Patients With Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-020
Record Dates: First submitted 2009-06-09; First posted 2009-06-26 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2013-04

CONDITIONS: Hypertension
Keywords: Hypertension; Resistant Hypertension; Sleep apnea syndrome; Treatment
MeSH Terms: conditions — Hypertension; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active CPAP (Active Comparator): auto-PAP with therapeutic pressure
  Interventions: Device: active CPAP
- sham-CPAP (Sham Comparator): auto-PAP with pressure less than 1cm H2O
  Interventions: Device: sham-CPAP

INTERVENTIONS:
Device: active CPAP — auto-PAP with pressure between 6 and 12 cm H2O or sham CPAP will be administered to randomized patients
  Arms: active CPAP
Device: sham-CPAP — The sham-CPAP was the same equipment used for active CPAP (Respironics Remstar-Auto, Murraysville, PA) fixed in the lowest pressure (4cmH2) and modified as recommended by Farré et al. The differences between the two were undetectable except for the pressure generated in the facial mask in the sham-CPAP that was no greater than 1cm H2O.
  Arms: sham-CPAP

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) has been linked to resistant hypertension, but the effect of treatment of OSAS on the resistant hypertension have no been established. In a double-blind randomized clinical trial patients with resistant hypertension with at least moderate sleep apnea will be randomized to receive therapeutic CPAP or Placebo CPAP for eight weeks in an ambulatory set. The investigators want to determine any difference on hypertension control between the 2 management strategies.

DETAILED DESCRIPTION:
This is a double blind, randomized, placebo controlled trial. Participants were consecutive patients with resistant hypertension, defined as uncontrolled BP, despite the concurrent use of 3 or more antihypertensive agents, including a diuretic, with adherence to treatment and without white coat phenomenon. All participants should have a diagnosis of at least moderate OSAS, defined by AHI > 15 in a portable monitoring sleep exam. Participants were assigned to active CPAP or sham-CPAP. The main outcome was change in 24-hour ambulatory blood pressure (ABP) monitoring values from baseline to two months of active CPAP or sham CPAP

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of resistant hypertension
* Apnea/hypopnea index > 15

Exclusion Criteria:

* Cardiac surgery on last 3 months
* Serious arrhythmias
* Insulin dependent diabetes
* Debilitating neurological disease
* severe COPD

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure evaluated with ambulatory 24-hour blood pressure monitoring | 8 weeks after treatment

SECONDARY OUTCOMES:
aldosterone, renin, activated protein C | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Flavio D Fuchs, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] de Oliveira AC, Martinez D, Massierer D, Gus M, Goncalves SC, Ghizzoni F, Steinhorst AM, Moreira LB, Fuchs SC, Fuchs FD. The antihypertensive effect of positive airway pressure on resistant hypertension of patients with obstructive sleep apnea: a randomized, double-blind, clinical trial. Am J Respir Crit Care Med. 2014 Aug 1;190(3):345-7. doi: 10.1164/rccm.201403-0479LE. No abstract available. PMID 25084263